CLINICAL TRIAL: NCT07096804
Title: Effects of Ramadan Fasting on Type 1 Diabetic Children in Assiut Governorate, Egypt
Brief Title: Effects of Ramadan Fasting on Type 1 Diabetic Children
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mahmoud Ismail Rashed, Resident Doctor, Assiut University
Other Study IDs: Diabetes and Ramadan fasting
Record Dates: First submitted 2025-07-22; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Diabtes Mellitus Type 1

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
assess the effects of Ramadan fasting on Type 1 diabetic children, fasting on their own, and to assess the validity of IDF-DAR risk calculator as a predictor of complications.

DETAILED DESCRIPTION:
Fasting during Ramadan holds profound religious, spiritual, and social significance for Muslims worldwide. This divine decree underscores the purpose of fasting, not merely as a physical exercise but as a means to develop spiritual consciousness and self-restraint. However, the Quran also provides allowances for those who are ill or incapable of fasting. This reflects Islam's principle of ḥifẓ al-nafs - the preservation of life, which takes precedence when health may be endangered . The practice of fasting during Ramadan entails abstaining from food, drink, medications, and other specific activities from dawn until sunset each day for a lunar month. For healthy adults, this fasting pattern generally carries spiritual and even certain metabolic benefits. However, for individuals with chronic diseases such as diabetes mellitus, particularly type 1 diabetes mellitus (T1DM) in children, fasting can present considerable challenges and potential dangers if not approached with caution and proper planning . The metabolic complexity of T1DM, especially in the pediatric population, demands careful medical and religious considerations before embarking on fasting .To guide healthcare professionals, the International Diabetes Federation (IDF) in collaboration with the Diabetes and Ramadan International Alliance (DaR) have developed comprehensive guidelines for managing patients with diabetes during Ramadan. The most critical component of these guidelines is a detailed risk stratification model, which categorizes patients into low, moderate, or high-risk groups based on various clinical factors . According to these guidelines, most children with T1DM - especially those with recent severe hypoglycemia, diabetic ketoacidosis, poor glycemic control, or limited access to monitoring technology - are classified as high-risk and are generally advised against fasting .Despite these risks, many children and families express a strong desire to participate in fasting as part of their religious practice. Studies have found that with appropriate preparation, some older children and adolescents with well-controlled T1DM could fast successfully without severe adverse events under close medical supervision . However, these studies also emphasized the importance of continuous glucose monitoring (CGM), flexible insulin regimens, and careful dietary planning to minimize glycemic excursions during fasting .Additionally, many children with type 1 diabetes in school settings express a strong desire to fast during Ramadan . This is often driven by a sense of embarrassment or peer pressure, as they do not want to appear different from their classmates. Religious motivation also plays a significant role, as these children wish to fulfill the spiritual obligation of fasting like their peers and family members .

ELIGIBILITY:
Inclusion Criteria: Children aged <18 years with established type 1 diabetes, on a stable insulin regimen (multiple daily injections or insulin pump) fasting Ramadan on their welling.

* Another comparable number of age and sex matched type 1 diabetic children not fasting will be included as a control.

Exclusion Criteria: patients with type 2 diabetes or seconadry diabetes

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with type 1 diabetes
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-02-25 (Estimated); Primary Completion 2028-02-25 (Estimated); Study Completion 2028-05-25 (Estimated)

PRIMARY OUTCOMES:
• Change in HbA1c from baseline to 4 weeks post-Ramadan. | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Hanaa Abdelateef Mohamad, Professor, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: No